CLINICAL TRIAL: NCT02204449
Title: Mentorship to Promote Cardiac Rehabilitation Enrollment: A Randomized Controlled Trial
Brief Title: Cardiac Rehabilitation Peer Mentorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Stony Brook University (Other); York University (Other)
Responsible Party: Principal Investigator, Sherry Grace, Full Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-7183
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Bypass Graft Surgery, With or Without Valve Surgery; Acute Coronary Syndrome; Chronic Stable Heart Failure; Coronary Artery Disease
Keywords: cardiac rehabilitation; peer mentorship; healthcare utilization; continuity of cardiac care
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiac Rehabilitation Peer Mentorship (Experimental): Trained cardiac rehabilitation (CR) peer mentors will visit cardiac inpatients in the hospital to provide patients with information on CR. During this visit the CR mentors will discuss the benefits of CR, stress the importance of getting a referral, and arrange a time to call the patient/participant at home to find out about their CR progress. One week post-discharge the peer mentor will mail a card to the patient to remind them of the planned call. Two weeks post-discharge the peer mentor will call the patient at home to determine if they were referred and if they are planning to attend CR. If any barriers are stated by patient the peer mentors will work with the patient to develop possible solutions. Patients can request up to two additional phone calls from the mentors.
  Interventions: Behavioral: Cardiac Rehabilitation Peer Mentorship
- Usual Care (No Intervention): Cardiac inpatients will not be visited by the cardiac rehabilitation (CR) peer mentor. They will instead receive usual care involving care from health care providers (i.e. nurses and doctors) as well as allied health professionals such as physiotherapists. In addition, some may be visited by general volunteer cardiac mentors.

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation Peer Mentorship
  Arms: Cardiac Rehabilitation Peer Mentorship

SUMMARY:
The current study is a randomized controlled trial, being conducted at two hospitals in Toronto, Ontario, Canada, involving the randomization of cardiac inpatients into an intervention group, in which they will receive mentorship from a volunteer cardiac rehabilitation peer mentor, and a control group, in which they will receive usual care. Patients in both groups will be tracked to determine if they are referred to cardiac rehabilitation and if they enroll in cardiac rehabilitation. We hypothesize that compared to cardiac inpatients who receive usual care, those cardiac inpatients who receive cardiac rehabilitation peer mentorship will be more likely to be referred to and enroll in cardiac rehabilitation.

DETAILED DESCRIPTION:
The current study will be a randomized controlled trial in which cardiac inpatients will be randomized to either receive the intervention (cardiac rehabilitation peer mentorship) or be in the control group (receive usual care). After consent is obtained cardiac patients in the intervention group will be visited, at the hospital bedside, by trained volunteer cardiac rehabilitation peer mentors (i.e., individuals who have completed cardiac rehabilitation) who will provide the patients with information on cardiac rehabilitation as well as encourage the patients to obtain a referral from their healthcare provider. During this visit the cardiac rehabilitation peer mentor will also obtain agreement from the patient to call the patient at home two weeks after their discharge. Those in the control group will not be visited by cardiac rehabilitation peer mentors.

One week after discharge the cardiac rehabilitation peer mentors will mail the patients in the intervention a get-well soon card reminding the patient of the visit, giving them more information about the cardiac rehabilitation program, and reminding them of their future scheduled phone call. Two weeks after patients' discharge cardiac rehabilitation peer mentors will call the patients in the intervention group. At this point they will assess how the patient is doing, if they were referred to cardiac rehabilitation and if they enrolled. Any possible barriers the patients have to attending cardiac rehabilitation will also be discussed.

Eight weeks post-discharge, patient referral and enrolment will be ascertained by a research assistant blinded to random assignment. Statistical analyses will be conducted to determine any differences between the two groups as well as to determine any differences between men and women.

ELIGIBILITY:
Inclusion Criteria:

* Any condition indicated for cardiac rehabilitation: Acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft +/- valve surgery or procedure (e.g., TAVI), heart transplant, ventricular assist device, heart failure, arrhythmia, rhythm device (i.e. implantable cardioverter-defibrillator, cardiac resynchronization therapy, pacemaker), congenital heart disease, minor non-disabling stroke or transient ischemic attack (i.e., can ambulate), peripheral vascular disease
* Proficiency in English language

Exclusion Criteria:

* Any musculoskeletal, neuromuscular, visual, cognitive or non-dysphoric psychiatric condition, or any serious or terminal illness not otherwise specified which would preclude CR eligibility based on CR guidelines
* Being discharged to long-term care
* Inability to ambulate (i.e. walk unaided at 2mph)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Grace, PhD, Principal Investigator — York University
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Ali-Faisal SF, Benz Scott L, Johnston L, Grace SL. Cardiac rehabilitation referral and enrolment across an academic health sciences centre with eReferral and peer navigation: a randomised controlled pilot trial. BMJ Open. 2016 Mar 21;6(3):e010214. doi: 10.1136/bmjopen-2015-010214. PMID 27000785

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Rehabilitation Peer Mentorship: Trained cardiac rehabilitation (CR) peer mentors will visit cardiac inpatients in the hospital to provide patients with information on CR. During this visit the CR mentors will discuss the benefits of CR, stress the importance of getting a referral before leaving the hospital, and arrange a time in the near future to call the patient/participant at home to find out about their progress in terms of CR.
  One week after the patient has been discharged the peer mentor will mail a card to the patient to wish them well and remind them of the planned call. Two weeks after the patient has been discharged the peer mentor will call the patient at home to determine if they were referred and if they are able and planning to attend CR. If any barriers are stated by the patient the peer mentors will work with the patient to develop possible solutions to those barriers. Patients can request up to two additional phone calls from the peer mentors.
  Cardiac Rehabilitation Peer Mentorship
Period: Overall Study
Arm/Group | Cardiac Rehabilitation Peer Mentorship | Usual Care
Started | 46 | 48
Completed | 39 | 37
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 7 | 9
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiac Rehabilitation Peer Mentorship | Usual Care | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (16.5) | 62.6 (13.1) | 62.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  Canada | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Rehabilitation Enrollment
Description: A blinded research assistant will either examine medical records or call the participant (i.e., patient) at home to determine if they have enrolled in cardiac rehabilitation.
Time Frame: 12 weeks after patient is discharged from hospital
Measure: Number; unit: participants
Arm/Group | Cardiac Rehabilitation Peer Mentorship | Usual Care
Number analyzed (Participants) | 39 | 37
participants | 20 | 15

2. Secondary Outcome: Cardiac Rehabilitation Referral
Description: A blinded research assistant will examine patient medical records to determine if patients were referred to cardiac rehabilitation.
Time Frame: 12 weeks after patient has been discharged from hospital
Measure: Number; unit: participants
Arm/Group | Cardiac Rehabilitation Peer Mentorship | Usual Care
Number analyzed (Participants) | 39 | 37
participants | 31 | 27

3. Other Pre Specified Outcome: Cardiac Rehabilitation Enrollment in Site Closer to Home
Description: A blinded research assistant will call those patients who were re-referred to a cardiac rehabilitation site closer to their home to see if they enrolled in cardiac rehabilitation. The study coordinator will then compare this to enrollment rates (already determined by the blinded research assistant) of those who enrolled in the program at the hospital system in which they were inpatients.
Time Frame: 8 weeks after patient is discharged from hospital
Measure: Number; unit: participants
Arm/Group | Cardiac Rehabilitation Peer Mentorship | Usual Care
Number analyzed (Participants) | 23 | 21
participants | 17 | 13

ADVERSE EVENTS:
Arm/Group | Cardiac Rehabilitation Peer Mentorship | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes